CLINICAL TRIAL: NCT00305357
Title: Evolution of Pain and Neural Dysfunction From Acute Herpes Zoster to Post-Herpetic Neuralgia
Brief Title: Evolution of Pain From Herpes Zoster
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Karin Petersen, MD, University of California, San Francisco
Other Study IDs: H5612-16138
Record Dates: First submitted 2006-03-17; First posted 2006-03-21 (Estimated); Last update posted 2023-05-24 (Actual); Status verified 2011-03

CONDITIONS: Post-Herpetic Neuralgia; Acute Herpes Zoster
Keywords: Post-Herpetic Neuralgia; Acute Herpes Zoster
MeSH Terms: conditions — Neuralgia, Postherpetic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Evolution of pain and neural injury will be evaluated at 2 years or longer after the onset of AHZ by multiple measures. Assessments at 2 years or longer will be compared to those collected during the first 6 months after HZ in order to test whether or not sensory function and cutaneous innervation continues to normalize beyond 6 months in subjects who recover from HZ without severe PHN.

DETAILED DESCRIPTION:
Pain, nerve trunk inflammation, and neuronal injury are hallmarks of acute herpes zoster (AHZ). We hypothesize that the development of post-herpetic neuralgia (PHN) strongly depends on two factors: 1) the severity of the initial neural injury and 2) the ability to recover from the initial neural injury. To test this hypothesis, we will prospectively follow 150 patients at high risk for development of PHN. Evolution of pain and neural injury will be evaluated at 2-6 weeks, 6 weeks, 3 months, 6 months and at 2 years or longer after the onset of AHZ by multiple measures. Assessments at 2 years or longer will be compared to those collected during the first 6 months after HZ in order to test whether or not sensory function and cutaneous innervation continues to normalize beyond 6 months in subjects who recover from HZ without severe PHN.

Preliminary analysis of study data showed reduced innervation in HZ skin, mirror image skin and distant control skin in the acute phase of HZ that was not specific to the persistence of pain at 3 months. The innervation appeared to recover more fully by 6 months in distant control skin than in mirror-image skin and HZ skin, despite the fact that the subjects were continuing to experience a further reduction in their zoster-associated pain. This suggests that the symptoms of pain and sensory dysfunction are not due to a mere loss in overall innervation density. The proposed subsequent ≥ 2 year study visit and analysis will allow us to directly correlate pain resolution with resolution of sensory and innervation abnormalities.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 50 or older and in stable general health.
2. Able and willing to provide written informed consent.
3. Able to understand and follow the instructions of the investigator, including the pain intensity rating scales.
4. Subjects must have an acute outbreak of cervical, thoracic or lumbosacral HZ with unilateral skin rash and pain; the diagnosis will be based on physical examination and review of available medical records confirming the outbreak.
5. The outbreak of herpes zoster must have occurred less than 6 weeks prior to study entry.
6. PHN pain must be of at least moderate severity, defined as self-report of average pain level of 20 mm on a 100 mm visual analog scale.

Exclusion Criteria:

1. The AHZ outbreak is complicated by stroke or myelopathy.
2. Patients with facial or cranial AHZ.
3. Patients with signs of spinal cord or brainstem injury from HZ.
4. Patients who are considered unreliable as to study compliance or adherence to scheduled appointments as determined by the Investigators.
5. Patients, who are undergoing active treatment for cancer, are infected with the Human Immunodeficiency Virus, or are being acutely and intensively immunosuppressed following a transplantation procedure.
6. Bleeding disorders.
7. Patients with known skin pathology.
8. Use of topical steroids, capsaicin, local anesthetics or topical aspirin/NSAID preparations within two weeks of the study sessions.
9. Another pain problem of equal or greater severity than AHZ.
10. Allergy or idiosyncratic reaction to lidocaine or capsaicin.
11. Neurological dysfunction or psychiatric disorder severe enough to interfere with assessment of pain and sensory systems.
12. Has received neuroablative nerve blocks or neurosurgical procedures for AHZ pain prior to entering the study.
13. Patients who are unable to read or speak English.
14. Those, in the opinion of the investigator, who are unlikely to comply with the study protocol or who are unsuitable for any other reason.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males and females aged 50 or older with outbreak of herpes zoster occurring less than 6 weeks prior to study entry.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2001-11; Primary Completion 2005-11 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karin Petersen, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF, San Francisco, California, United States